CLINICAL TRIAL: NCT00081731
Title: Cardiovascular Outcomes in Renal Atherosclerotic Lesions (CORAL)
Brief Title: Benefits of Medical Therapy Plus Stenting for Renal Atherosclerotic Lesions
Acronym: CORAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 161; U01HL071556 (NIH)
Record Dates: First submitted 2004-04-19; First posted 2004-04-21 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Hypertension, Renovascular; Renal Artery Obstruction
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Hypertension, Renovascular; Renal Artery Obstruction | interventions — amlodipine, atorvastatin drug combination; Angioplasty; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal Medical Therapy (Active Comparator): Optimal anti-hypertensive therapy
  Interventions: Drug: Atacand/HCT, Caduet
- Stenting (Experimental): Stent procedure plus optimal anti-hypertensive therapy
  Interventions: Procedure: GENESISTM Embolic Protection Stent and Angioguard Device (Angioplasty plus stenting)

INTERVENTIONS:
Drug: Atacand/HCT, Caduet — Atacand/HCT and caduet or optimal medical therapy for hypertension
  Arms: Optimal Medical Therapy
Procedure: GENESISTM Embolic Protection Stent and Angioguard Device (Angioplasty plus stenting) — Angioplasty plus stenting of the renal artery GENESISTM Embolic Protection Stent and Angioguard Device
  Arms: Stenting

SUMMARY:
This study will compare medical therapy plus stenting of hemodynamically significant renal artery stenoses versus medical therapy alone in patients with systolic hypertension and renal artery stenosis.

DETAILED DESCRIPTION:
BACKGROUND:

Atherosclerotic renal artery stenosis is a common problem for which there is no clear consensus on diagnosis or therapy. There likely exists a progression in which renal ischemia leads to neuroendocrine activation, hypertension, and renal insufficiency resulting in acceleration of atherosclerosis, further renal dysfunction, and development of left ventricular hypertrophy. These events in turn lead to adverse clinical events.

Renal artery stenosis is one of the two major known causes of hypertension and occurs in 1-5% of hypertensive patients. In patients with accelerated hypertension, the prevalence of renal artery stenosis is much higher, ranging from 10-40%. Renal artery stenosis, when occurring bilaterally, or in a solitary kidney, is a significant cause for end-stage renal disease, accounting for several percent of patients with end-stage renal disease. Clinically, atherosclerotic renal artery stenosis is a major problem primarily in older patients, and is often seen in long-standing hypertensives whose blood pressure becomes very difficult to control. Of major significance is the progressive nature of atherosclerotic renal artery stenosis, progressing at the rate of about 10% per year (45-60% progression rate in 4-7 year follow-ups). Over this time period, 10-15% of patients develop total renal artery occlusion. If the renal artery stenosis is greater than 75% when detected, 40% of patients develop total occlusion. Due to the progressive nature of atherosclerotic lesions, the decline in renal function in some individuals, and difficult-to-control hypertension, the medical community has sought to detect those patients in whom intervention would be beneficial. This has been extremely difficult to achieve and tests to date have not been uniformly predictive, including peripheral vein plasma renin activity, renal vein renin activity, captopril-stimulated nuclear medicine renal scans, etc.

Since approximately 50% of patients with unilateral renal artery stenosis of significant degree (definitions vary) benefit from surgical intervention, enthusiasm has continued with the advent of renal artery angioplasty. The entire field is moving very quickly. However, there are neither current data nor prospective studies indicating the benefit of renal artery angioplasty plus stents. Studies over the last decade have shown that balloon angioplasty alone is associated with a high rate of recurrence in patients with atherosclerotic renal artery stenosis. In the present climate, there is great enthusiasm to perform angioplasty plus stent placement in atherosclerotic renal artery stenosis, without supporting data for efficacy compared to medical management alone. Angioplasty and stent placement in the renal arteries had been the domain of interventional radiologists, but recently, interventional cardiologists are also performing these procedures. The questions as to who will benefit from intervention and which intervention to use have not been answered. Renal artery angioplasty and stent placement subjects the patient to procedural risks, as well as increased cost, when compared to aggressive antihypertensive medication and risk factor medication and therapy.

DESIGN NARRATIVE:

This randomized, multicenter clinical trial will contrast the effect of optimal medical therapy alone to stenting with optimal medical therapy, on a composite of cardiovascular and renal endpoints: cardiovascular or renal death, myocardial infarction, hospitalization for congestive heart failure, stroke, doubling of serum creatinine level, and need for renal replacement therapy. These endpoints will be evaluated by a clinical events committee masked to treatment assignment. The secondary endpoints will 1) evaluate the mechanisms linked to clinical events; 2) describe differential effectiveness in critical end-organs; 3) determine the value of stenting from the patient and the health policy perspectives, measured as quality of life and cost-effectiveness; and 4) evaluate for clinically relevant differences in treatment effectiveness within the primary endpoint.

Patients will undergo a baseline evaluation to determine eligibility. Approximately 1,080 patients will be randomized to optimal medical therapy alone or to stenting with optimal medical therapy at an estimated 100 clinical sites. Initially, patients will be followed at 2-week intervals, until blood pressure is at target or up to 2 months. Follow-up visits will be mandated at 2 weeks, every 3 months for the first year and annually thereafter. Coordinator visits will also occur semi-annually.

The CORAL Study Chair is Lance Dworkin, MD, Brown University, Providence, RI. The CORAL Study Co-Chair is William Henrich, MD, University of Texas, San Antonio, TX. The Principal Investigators of the CORAL Clinical Coordinating Center are Christopher Cooper, MD, University of Toledo Health Science Campus, Toledo OH, and Timothy Murphy, MD, Brown University, Providence, RI.

The Principal Investigator of the Angiographic Core Laboratory is Alan Matsumoto, MD, University of Virginia, Charlottesville, VA. The Principal Investigator of the GFR and Biochemistry Core Laboratory is Michael Steffes, MD, University of Minnesota, Minneapolis, MN. The Principal Investigator of the Economics and Quality of Life Core Laboratory is David Cohen, MD, Mid-America Heart Institute, St. Luke's Hospital, Kansas City, MO. The Principal Investigator of the Data Coordinating Center is Donald Cutlip, MD, Beth Israel Deaconess Medical Center, Boston, MA. For additional information about the CORAL trial, please refer to the CORAL website (link given below).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Either

   1. Documented history of hypertension on two or more anti-hypertensive medications OR
   2. Renal dysfunction, defined as Stage 3 or greater chronic kidney disease (CKD) based on the new National Kidney Foundation (NKF) classifications (estimated glomerular filtration rate [GFR] less than 60 mL per minute per 1.73 m^2, calculated by the modified Modification of Diet in Renal Disease [MDRD] formula)
2. One or more severe renal artery stenoses by any of the following pathways:

   a. Angiographic: greater than or equal to 60% and less than 100% by renal angiogram OR b. Duplex: systolic velocity of greater than 300 cm/sec OR c. Core Lab approved Magnetic Resonance Angiogram (MRA) (refer to the protocol for specific criteria) demonstrating stenosis greater than 80% OR stenosis greater than 70% with spin dephasing on 3D phase contrast MRA OR stenosis greater than 70% and two of the following: i. Ischemic kidney is greater than 1 cm. smaller than contralateral kidney ii. Ischemic kidney enhances less on arterial phase iii. Ischemic kidney has delayed Gd excretion iv. Ischemic kidney hyper-concentrates the urine v. 2-D phase contrast flow waveform shows delayed systolic peak vi. Post-stenotic dilatation d. Clinical index of suspicion combined with a Core Lab approved Computed Tomography Angiography (CTA) demonstrating Stenosis is greater than 80% by visual assessment on high quality CTA Stenosis is greater than 70% on CTA by visual assessment and there are two of the following i. The length of the ischemic kidney is greater than 1 cm. smaller than contralateral kidney ii. Reduced cortical thickness of ischemic kidney iii. Less cortical enhancement of ischemic kidney on arterial phase iv. Post-stenotic dilatation

EXCLUSION CRITERIA:

1. Unable to provide informed consent
2. Unable or willing to comply with study protocol or procedures
3. Must be greater than 18 years of age
4. Fibromuscular dysplasia or other non-atherosclerotic renal artery stenosis known to be present prior to randomization
5. Pregnancy or unknown pregnancy status in female of childbearing potential
6. Participation in any drug or device trial during the study period, unless approved by the Steering Committee
7. Prior enrollment in the CORAL study
8. History of stroke within 6 months, if associated with a residual neurologic deficit*
9. Any major surgery, major trauma, revascularization procedure, unstable angina, or myocardial infarction 30 days prior to study entry*
10. Any planned major surgery or revascularization procedure, outside of the randomly allocated renal stenting indicated by the protocol, after randomization*
11. Hospitalization for heart failure within 30 days*
12. Comorbid condition causing life expectancy of less than or equal to 3 years*
13. Allergic reaction to intravascular contrast, not amenable to pre-treatment
14. Allergy to stainless steel
15. Allergy to all of the following: aspirin, clopidogrel, ticlopidine
16. Known untreated aneurysm of the abdominal aorta greater than 5.0 cm.*
17. Previous kidney transplant
18. a. Stenosis of greater than 50% of a previously treated revascularized renal artery OR b. Treatment of any renal artery stenosis within the past 9 months (roll-in patients can have prior treatment on the contralateral side)
19. Kidney size less than 7 cm. supplied by target vessel
20. Hydronephrosis, nephritis or other known cause of renal insufficiency, not due to large vessel renal artery stenosis
21. Visualized stenosis of only an accessory renal artery supplying greater than 1/2 of the ipsilateral renal parenchyma, without stenosis in a dominant renal artery
22. Local lab serum Cr greater than 4.0 mg/dl on the day of randomization*
23. Presence of a renal artery stenosis not amenable for treatment with a stent, known to be present prior to randomization

    1. The index lesion cannot be treated with a single stent (i.e. greater than 18 mm. in length)
    2. The placement of a stent will necessitate covering a renal artery branch renal artery with a stent
    3. The stenosis is in an artery less than 3.5 mm. in diameter
    4. The stenosis involves a segmental renal artery branch
24. Abrupt vessel closure or dissection after diagnostic angiography [NOTE: Patients with abrupt vessel closure or dissection as a result of diagnostic angiography will not be randomized but will undergo stent revascularization, receive optimal medical therapy and will be followed for the full study period] *Roll-in patients do not need to meet these inclusion/exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2004-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cohen, MD, Principal Investigator — Mid-America Heart Institute, St. Luke's Hospital, Kansas City, MO; Christopher J. Cooper, MD, Principal Investigator — University of Toledo; Donald Cutlip, MD, Principal Investigator — Beth Israel Deaconess Medcial Center; Alan Matsumoto, MD, Principal Investigator — University of Virginia School of Medicine; Michael Steffes, MD, Principal Investigator — University of Minnesota; Timothy P Murphy, MD, Principal Investigator — Rhode Island Hospital; Scott D Solomon, MD, Study Chair — Brigham and Women's Hospital; Lance D Dworkin, MD, Study Chair — Rhode Island Hospital
Locations (1):
- University of Toledo, Toledo, Ohio, United States

REFERENCES:
- [Background] Cooper CJ, Murphy TP, Matsumoto A, Steffes M, Cohen DJ, Jaff M, Kuntz R, Jamerson K, Reid D, Rosenfield K, Rundback J, D'Agostino R, Henrich W, Dworkin L. Stent revascularization for the prevention of cardiovascular and renal events among patients with renal artery stenosis and systolic hypertension: rationale and design of the CORAL trial. Am Heart J. 2006 Jul;152(1):59-66. doi: 10.1016/j.ahj.2005.09.011. PMID 16824832
- [Background] Murphy TP, Cooper CJ, Dworkin LD, Henrich WL, Rundback JH, Matsumoto AH, Jamerson KA, D'Agostino RB. The Cardiovascular Outcomes with Renal Atherosclerotic Lesions (CORAL) study: rationale and methods. J Vasc Interv Radiol. 2005 Oct;16(10):1295-300. doi: 10.1097/01.RVI.0000176301.69756.28. No abstract available. PMID 16221898
- [Result] Bittl JA. Treatment of atherosclerotic renovascular disease. N Engl J Med. 2014 Jan 2;370(1):78-9. doi: 10.1056/NEJMe1313423. Epub 2013 Nov 18. No abstract available. PMID 24245567
- [Derived] Arnold SV, Wang K, Kirtane AJ, Magnuson EA, Chinnakondepalli KM, Cooper CJ, Dworkin LD, Cohen DJ. Quality of life effects of renal artery stenting versus medical therapy for atherosclerotic renal-artery stenosis: results from the randomized CORAL trial. Eur Heart J Qual Care Clin Outcomes. 2025 Dec 19;11(8):1388-1395. doi: 10.1093/ehjqcco/qcae087. PMID 39402005
- [Derived] Lerman LO. Cell-based regenerative medicine for renovascular disease. Trends Mol Med. 2021 Sep;27(9):882-894. doi: 10.1016/j.molmed.2021.06.004. Epub 2021 Jun 25. PMID 34183258
- [Derived] Chen T, Brewster P, Tuttle KR, Dworkin LD, Henrich W, Greco BA, Steffes M, Tobe S, Jamerson K, Pencina K, Massaro JM, D'Agostino RB Sr, Cutlip DE, Murphy TP, Cooper CJ, Shapiro JI. Prediction of cardiovascular outcomes with machine learning techniques: application to the Cardiovascular Outcomes in Renal Atherosclerotic Lesions (CORAL) study. Int J Nephrol Renovasc Dis. 2019 Mar 21;12:49-58. doi: 10.2147/IJNRD.S194727. eCollection 2019. PMID 30962703
- [Derived] Murphy TP, Cooper CJ, Pencina KM, D'Agostino R, Massaro J, Cutlip DE, Jamerson K, Matsumoto AH, Henrich W, Shapiro JI, Tuttle KR, Cohen DJ, Steffes M, Gao Q, Metzger DC, Abernethy WB, Textor SC, Briguglio J, Hirsch AT, Tobe S, Dworkin LD. Relationship of Albuminuria and Renal Artery Stent Outcomes: Results From the CORAL Randomized Clinical Trial (Cardiovascular Outcomes With Renal Artery Lesions). Hypertension. 2016 Nov;68(5):1145-1152. doi: 10.1161/HYPERTENSIONAHA.116.07744. Epub 2016 Sep 19. PMID 27647847
- [Derived] Murphy TP, Cooper CJ, Matsumoto AH, Cutlip DE, Pencina KM, Jamerson K, Tuttle KR, Shapiro JI, D'Agostino R, Massaro J, Henrich W, Dworkin LD. Renal Artery Stent Outcomes: Effect of Baseline Blood Pressure, Stenosis Severity, and Translesion Pressure Gradient. J Am Coll Cardiol. 2015 Dec 8;66(22):2487-94. doi: 10.1016/j.jacc.2015.09.073. PMID 26653621
- [Derived] Evans KL, Tuttle KR, Folt DA, Dawson T, Haller ST, Brewster PS, He W, Jamerson K, Dworkin LD, Cutlip DE, Murphy TP, D'Agostino RB Sr, Henrich W, Cooper CJ. Use of renin-angiotensin inhibitors in people with renal artery stenosis. Clin J Am Soc Nephrol. 2014 Jul;9(7):1199-206. doi: 10.2215/CJN.11611113. Epub 2014 Jun 5. PMID 24903387
- [Derived] Murphy TP, Cooper CJ, Cutlip DE, Matsumoto A, Jamerson K, Rundback J, Rosenfield KA, Henrich W, Shapiro J, Massaro J, Yen CH, Burtch H, Thum C, Reid D, Dworkin L. Roll-in experience from the Cardiovascular Outcomes with Renal Atherosclerotic Lesions (CORAL) study. J Vasc Interv Radiol. 2014 Apr;25(4):511-20. doi: 10.1016/j.jvir.2013.09.018. Epub 2013 Dec 8. PMID 24325931
- [Derived] Cooper CJ, Murphy TP, Cutlip DE, Jamerson K, Henrich W, Reid DM, Cohen DJ, Matsumoto AH, Steffes M, Jaff MR, Prince MR, Lewis EF, Tuttle KR, Shapiro JI, Rundback JH, Massaro JM, D'Agostino RB Sr, Dworkin LD; CORAL Investigators. Stenting and medical therapy for atherosclerotic renal-artery stenosis. N Engl J Med. 2014 Jan 2;370(1):13-22. doi: 10.1056/NEJMoa1310753. Epub 2013 Nov 18. PMID 24245566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optimal Medical Therapy | Stenting
Started | 480 | 467
Completed | 472 | 459
Not Completed | 8 | 8
Not completed — scientific integrity issue | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimal Medical Therapy | Stenting | Total
Number analyzed (Participants) | 472 | 459 | 931
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9.0) | 69.3 (9.4) | 69.15 (9.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 140 | 127 | 267
  >=65 years | 332 | 332 | 664
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 225 | 466
  Male | 231 | 234 | 465
Region of Enrollment [Number; unit: participants]
  United States | 387 | 385 | 772

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint: Death From Cardiovascular or Renal Causes, Stroke, Myocardial Infarction, Hospitalization for CHF, Progressive Renal Insufficiency, or Permanent Renal Replacement Therapy
Description: Only the first event per participant is included in the composite
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 169 [0.76 to 1.17] | 161 [0.76 to 1.17]

2. Primary Outcome: Cardiovascular or Renal Death
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 20 | 20

3. Primary Outcome: Myocardial Infarction
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 27 | 30

4. Primary Outcome: Hospitalization for Congestive Heart Failure
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 26 | 27

5. Primary Outcome: Stroke
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 16 | 12

6. Primary Outcome: 30% Reduction of eGFR From Baseline, Persisting for Greater Than or Equal to 60 Days
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 77 | 68

7. Primary Outcome: Need for Renal Replacement Therapy
Time Frame: Measured at every 3 months for the first year and annually thereafter
Measure: Number; unit: participants
Arm/Group | Optimal Medical Therapy | Stenting
Number analyzed (Participants) | 472 | 459
participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | Optimal Medical Therapy | Stenting
Serious Adverse Events (participants affected / at risk) | 283/472 | 290/459
Other Adverse Events (participants affected / at risk) | 441/472 | 429/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Medical Therapy (N=472) | Stenting (N=459)
Cardiac Disorders (Cardiac disorders) | 117 (117) | 128 (128)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 11 (11) | 16 (16)
Congenital, Familial and Genetic Disorders (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Eye Disorders (Eye disorders) | 3 (3) | 2 (2)
Gastrointestinal Disorders (Gastrointestinal disorders) | 42 (42) | 57 (57)
General Disorders (General disorders) | 38 (38) | 36 (36)
Hepatobiliary Disorders (Hepatobiliary disorders) | 7 (7) | 5 (5)
Immune System Disorders (Immune system disorders) | 0 (0) | 1 (1)
Infections and Infestations (Infections and infestations) | 69 (69) | 63 (63)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 19 (19) | 42 (42)
Investigations (Investigations) | 1 (1) | 4 (4)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 28 (28) | 19 (19)
Musuloskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 31 (31) | 39 (39)
Neoplasms Benign, Malignant and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 (26) | 27 (27)
Nervous System Disorders (Nervous system disorders) | 67 (67) | 61 (61)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Medical Therapy (N=472) | Stenting (N=459)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 93 (93) | 85 (85)
Cardiac Disorders (Cardiac disorders) | 205 (205) | 201 (201)
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 24 (24) | 32 (32)
Eye Disorders (Eye disorders) | 63 (63) | 60 (60)
General Disorders (General disorders) | 261 (261) | 251 (251)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 122 (122) | 133 (133)
Investigations (Investigations) | 125 (125) | 124 (124)

LIMITATIONS AND CAVEATS:
Patients could be enrolled in the trial with renal artery stenosis > = 60%. Didn't include patients with fibromuscular dysplasia. Some screened and deemed to be eligible were not enrolled because of physician preference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No